CLINICAL TRIAL: NCT05275816
Title: Appropriateness of Carpal Tunnel Syndrome Management Compared With the AAOS Appropriate Use Criteria: A Retrospective Review Across Various Specialties
Brief Title: Appropriateness of Carpal Tunnel Syndrome Management Compared With the AAOS Appropriate Use Criteria
Acronym: CTS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MRC-01-22-085
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal tunnel syndrome; Management; Hand Surgery
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Comparing the appropriateness of our practice and the usability of the AUC through comparing the actual management provided at our institution with that recommended by the AUC. — The AUC application for carpal tunnel syndrome management requires four patients' variables to generate appropriateness ratings for six different treatment options. Each procedure is rated as appropriate, maybe appropriate, or rarely appropriate. The six procedures include splint, steroid injection, carpal tunnel release, oral steroids or Ketoprofen phonophoresis, investigation of alternative diagnoses, and further investigation using an electro-diagnostic study.
  To judge the usability of the AUC for the management of carpal tunnel syndrome, the required parameters of each patient were collected and entered into the AUC application by two independent authors to generate the appropriateness rating of the provided treatment for each patient. Afterwards, the agreement between the AUC recommendations and the actual treatment that was provided at our institution was assessed.

SUMMARY:
Purpose: Carpal tunnel syndrome (CTS) is a common peripheral nerve entrapment disorder among adults that causes upper-extremity disability. The American Academy of Orthopedic Surgeons (AAOS) developed an evidence-based appropriate use criteria (AUC) for the management of CTS. This study aims to assess the appropriateness of our practice and the usability of the AUC by comparing the actual management provided at our institution with that recommended by the AUC.

Methods: A retrospective review of the electronic medical records at our hospital will be performed between 1 Jan 2016 and 31 Dec 2019. Data will be collected by two authors independently. The collected data will be input into the AUC application to determine the rate of the appropriateness of the treatments. Afterwards, the agreement between the actual treatment provided and the AUC recommendation will be assessed. The primary outcome will be the appropriateness rate. Descriptive statistics such as the mean, range and percentage will be used to summarize the patients' demographics and treatment options.

Results: The appropriateness rating (appropriate, maybe, or rarely appropriate) for each treatment will be described with percentages. Similarly, the agreement of the treatments implemented at our institution with the AUC recommendations will be expressed as a proportion. A subgroup analysis within the same cohort compared the appropriateness rates of surgical release of patients across different surgical specialties using chi2 test.

Conclusion: This study will show if the management provided at our institution were appropriate and in agreement with the AUC recommendations. Additionally, it will test the usability of AUC for carpal tunnel syndrome as a valuable and practical tool that can be applied in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years) who were diagnosed with CTS.

Exclusion Criteria as per the AUC:

* Acute carpal tunnel syndrome
* Untreated inflammatory arthritis
* Untreated diabetes
* Thyroid disease
* Pernicious Anemia
* Patients with a known space-occupying lesion in the carpal tunnel
* Failed treatment after surgery
* Pediatric and adolescent patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients presented to HGH or Bone and Joint Center and were diagnosed with carpal tunnel syndrome.
  Patients will be selected from computer-based case logs of HGH and Bone and Joint Centre in Doha, Qatar. The eligibility criteria were according to the AUC criteria for CTS management in adults.
Sampling Method: Probability Sample
Enrollment: 136 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
The rate of appropriateness of CTS management in our practice compared to the AUC recommendation | 4 months
  AUC Appropriateness rate (percentage/Continuous outcome): The AUC application for carpal tunnel syndrome management requires four patients' variables to generate appropriateness ratings for six different treatment options. Each procedure is rated as appropriate, maybe appropriate, or rarely appropriate. The six procedures include splint, steroid injection, carpal tunnel release, oral steroids or Ketoprofen phonophoresis, investigation of alternative diagnoses, and further investigation using an electro-diagnostic study.
  To judge the appropriateness of the AUC for the management of carpal tunnel syndrome, the required parameters of each patient were collected and entered into the AUC application by two independent authors to generate the appropriateness rating of the provided treatment for each patient. Afterwards, the agreement between the AUC recommendations and the actual treatment that was provided at our institution was assessed.

IPD SHARING:
Plan to Share IPD: Undecided